CLINICAL TRIAL: NCT04438629
Title: Evaluation of Immune Response in COVID-19 Patients
Acronym: IMMUNOVID
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Responsible Party: Sponsor
Other Study IDs: IMMUNOVID 2590CESC
Record Dates: First submitted 2020-06-16; First posted 2020-06-19 (Actual); Last update posted 2020-06-22 (Actual); Status verified 2020-03

CONDITIONS: Allergy and Immunology; Infection Viral
Keywords: COVID-19; IMMUNE SYSTEM; INNATE IMMUNITY; ADAPTIVE IMMUNITY
MeSH Terms: conditions — Hypersensitivity; Virus Diseases; COVID-19 | interventions — COVID-19 Drug Treatment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Mild disease: COVID-19 hospitalized patients
  Interventions: Drug: COVID-19 treatment
- Severe disease: COVID-19 hospitalized patients in intensive care unit
  Interventions: Drug: COVID-19 treatment
- paucisymptomatic syndrome: Mild symptomatic patients in home quarantine
  Interventions: Drug: COVID-19 treatment

INTERVENTIONS:
Drug: COVID-19 treatment — COVID-19 affected patients treated with hydroxicloroquine or antiviral therapy (lopinavir/ritonavir) as single agents or in combination (hydroxicloroquine plus antiviral therapy) according to clinical features. Other concomitant treatments (i.e. off-label therapy) will be provided at the discretion of clinicians. Supportive therapy, such as antibiotic prophylaxis and anticoagulant treatment, will be provided at the discretion of the clinicians.

SUMMARY:
The aim of the project is to evaluate the immunological features of COVID-19 patients. Patients are recruited without any pharmacological treatments restriction. The number of samples is estimated on the basis of feasibility, that means on the maximum number of patients with COVID-19, who are expected to be able to be enrolled by the units involved. Based on the investigators' experience, gained in the onco-immunological field, considering the time and economic resources available, the investigators expect to enroll at least 80 patients.

DETAILED DESCRIPTION:
PURPOSES

1. Determine the frequency of circulating immune cells (i.e. T cells, B cells, Neutrophils, Monocytes absolute numbers) in COVID-19 patients at Hospital Trust of Verona.
2. Determine the plasma levels of soluble factors (i.e. IL-1beta, IL-6, IL-10, TNFalfa) in COVID-19 patients at Hospital Trust of Verona.
3. Determinate the immune composition of lung and blood of COVID-19 patients that will be enrolled at Hospital Trust of Verona through single-cell sequencing analysis, capable of detecting also the viral sequences in each leukocyte populations.
4. Determine any potential links between cytokine storm, immune cells composition and clinical parameters (i.e.) in COVID-19 patients
5. Profile patients with a different stage of disease to identify potential biomarkers
6. Identify SARS-CoV-2-associated sequences in immune cells
7. To define differences in immune cell composition the immune profiling will be done before and after patients treatment used as part of clinical care in COVID-19 patients.

HYPOTHESES

1. Primary: Based on previous reports, COVID-19 patients showed significant immunological alterations that need to be deeply investigated. Therefore, the main objective of this study is to perform a phenotypic characterization of patients with COVID-19
2. Secondary: Immunological disorder induced by the infection can generate a systemic pathology. Therefore, a) the investigators will identify potential immune-associated biomarkers for rapid testing; b) the investigators will identify specific viral sequences inside immune cells that can explain the systemic disease c) the investigators will define immunological parameters that correlate with disease progression

JUSTIFICATION

The pandemic spread of a novel, highly pathogenic coronavirus (SARS-CoV-2) has found the international medical community largely unprepared on prophylactic and therapeutic measures. The resulting syndrome, known as COVID-19, is characterized by a profound dysfunction of the upper and lower respiratory tract, with severity ranging from mild to moderate respiratory failure, up to acute respiratory distress syndrome (ARDS) that is generally fatal2. Recently, the crucial role of the "cytokine release syndrome (CRS), also referred to as "cytokine storm", in acute lung damage and ARDS4,5 has become evident, thus providing the theoretical ground for therapeutic approaches able to interfere with the inflammatory cascade. Indeed, while the majority of patients either asymptomatic or with early stage of the disease are able to clear the infection, some patients with moderate disease, requiring hospital admittance, progress to a clinically severe phase associated with the "cytokine storm" within 10 days from symptom onset.

Delineation of a link between clinical parameters and immunological profile would provide a rational to define the perfect treatment to reduce the incidence of COVID-19 associated ARDS and mortality.

OBJECTIVES

Better understand 1) the link between immunological modifications and ARDS in COVID-19 patients; 2) the biomarker profile of COVID-19 patients with mild and severe disease; 3) the impact of virus sequences in circulating immune cells on clinical outcomes in COVID-19 patients

RESEARCH DESIGN

Patients admitted to Hospital Trust of Verona will be isolated in Infective Unit or intensive care unit (ICU) on basis of the . Here, specimens will be collected for laboratory confirmation of SARS-CoV-2 using nasopharyngeal swab assessed PCR by the Microbiology and Virology Unit. Clinical care will commence following the discretion of attending physicians in accordance with Hospital Trust of Verona current operating procedures for the management of COVID-19.

Once clinical care has commenced, a blood sample will be collected in three different moments: T0 = at diagnosis (which is equivalent for severe symptoms that will begin a therapeutic course, or for light symptoms within 72 hours from the COVID-19 diagnosis) ; T 1= after 7 days from diagnosis (for patients admitted to the UOC the collection will be carried out at the Operative Unit while for asymptomatic patients this collection will be done at the patient's home by health workers and then the sample will be sent to the Immunology Section); T2 = after 14 days from diagnosis similar to that described for the previous collection. All the samples will be collected into vacutainer serum separator tubes (SST, Vacutainer®, Becton & Dickinson). In some cases, patients admitted to ICU also receive BAL (bronchiole-alveolar lavage) or tracheal / mini BAL aspiration. The BAL will be collected whenever it is an integral part of the patient's diagnostic path or within thirty minutes of the patient's confirmed death. In all cases, together with the BAL it will also be necessary to collect a test tube of blood, independently and in addition to the samples described above.

These samples will be analyzed for: a) a complete immune phenotype by flow cytometry; b) a panel of soluble factots (i.e. cytokines), c) a deep immunological composition by single-cell RNA sequencing, d) presence of viral sequences.

Analysis will be performed at Immunology Section (a,b,c) and Microbiology and Virology Section of Hospital Trust of Verona.

Immunophenotype analysis on whole peripheral blood will be performed according to a standard no-wash procedure, using a PrepPlus™ 2 workstation (Beckman Coulter Inc., Brea, CA, USA). Blood samples will be incubated with antibodies (Beckman Coulter Inc., Brea, CA, USA) for 15 min at 20°C. Following is the list of antibodies used:

* FITC-conjugated CD57 (clone NC1), PE-conjugated CD45RA (ALB11), ECD-conjugated CD8 (SFCI21Thy2D3), PC5.5-conjugated CD56 (N901), PC7-conjugated CD4 (SFCI12T4D11), APC-conjugated CD27 (1A4CD27), APC A700-conjugated CD45 (J33), APC A750-conjugated CD3 (UCHT1), PB-conjugated CD16 (3G8), KR OR-conjugated CD19 (J3-119)
* FITC-conjugated CD57 (clone NC1), PE-conjugated HLA-DR (Immu-357), ECD-conjugated CD8 (SFCI21Thy2D3), PC5.5-conjugated CD38 (LS198-4-3), PC7-conjugated CD4 (clone SFCI12T4D11), APC-conjugated CD14 (RMO52), APC A700-conjugated CD45 (J33), APC A750-conjugated CD3 (UCHT1), PB-conjugated CD16 (3G8), KR OR-conjugated CD19 (J3-119)
* PE-conjugated IgD (IA6-2), ECD-conjugated CD3 (UCHT1), PC5.5-conjugated CD27 (1A4CD27), PC7-conjugated CD20 (clone B9E9), APC-conjugated IgM (SA-DA4), APC A700-conjugated CD45 (J33), APC A750-conjugated CD38 (LS198-4-3), PB-conjugated CD21 (BL13), KR OR-conjugated CD19 (J3-119) Red blood cell lysis and cell fixation will be performed using TQ-Prep workstation and ImmunoPrep reagent system (Beckman Coulter Inc., Brea, CA, USA). Samples will be acquired with Navios and analyzed with Navios software (Beckman Coulter Inc., Brea, CA, USA).

For detection of cytokines, sera of COVID-19 patients were tested for GM-CSF, G-CSF, M-CSF, IFN-γ, IFN-α, IL-1, IL-2, IL-4, IL-5, IL-6, IL-9, IL-10, IL-12 (p70), IL-13, IL-15, IL-17A, IL-17F, IL-17E, IL-21, IL-22, IL-23, IL-27, IL-28A, IL-31, IL-33, IL-34, MIP-3α/CCL20, CCL2, TNF-α, TNF-β, TGFβ production by Human ProcartaPlex™ Panel 1 multiplex (ThermoFisher Scientific, Waltham, MA, USA).

BAL cells and circulating immune cells will be purified and cell counts will be adjusted following 10xgenomics protocol. Briefly, the cell suspension was super-loaded with 50,000 cells, in the ChromiumTM Controller for partitioning single cells into nanoliter-scale Gel Bead-In-Emulsions (GEMs). Single Cell 3' reagent kit v3.1 will be used for reverse transcription, cDNA amplification and library construction of the gene expression libraries (10x Genomics) following the detailed protocol provided by 10xGenomics. Hashtag libraries will be prepared according to the cell hashing protocol for 10x Single Cell 3' Reagent Kit v3.1. Biometra Trio Thermal Cycler will be used for amplification and incubation steps (Analytik Jena). Libraries will be quantified by QubitTM 2.0 Fluorometer (ThermoFisher) and quality will be checked using 2100 Bioanalyzer with High Sensitivity DNA kit (Agilent). Sequencing will be performed in paired-end mode with a S1 and S2 flow cell (2 × 50 cycles kit) using NovaSeq 6000 sequencer (Illumina).

The short history of this disease outbreak makes robust statistical power testing difficult. However, for analysis during the treatment the investigators will consider only those patients who are still alive, for whom the clinical and laboratory data for at least two time points are available. Analysis on the duration of hospitalization will be performed in all the patients enrolled except for the ones who died. Quantitative variables will be expressed as the median and interquartile range (IQR), qualitative ones as percentages. To perform pairwise comparisons, significance of difference will be evaluated by the Mann-Witney U-test for quantitative variables and Fisher's exact test for categorical variables. The Wilcoxon matched-pairs signed-rank test will be used to test the equality of matched pairs of observation. Multiple logistic-regression analysis will be performed to assess the association between the treatment and mortality for known negative prognostic factor (age, sex and D-dimer). The strength of the association will be expressed by the Hazard Ratio (HR) with 95% confidence interval (CI). Statistical significance will set at p-value <0.05, and clinical analyses will be performed using statistical software STATA version 16.0 (StataCorp, College Station, TX, USA). For statistical laboratory analyses the investigators will perform paired comparisons by Student's t-test and one-way Anova test for repeated measures, using Graph Pad Prism (San Diego, California, version 8.4.2).

All biological materials will be stored after anonymisation at of Medicine Department of University and Hospital Trust of Verona for the duration of the study (8 months). After that, all biological materials will be transferred at Biobanca of University and Hospital Trust of Verona. All patients data will be only accessed by researchers involved in the study with a personnel account. All patients are anonymzed during immunological analysis. All data are protected by software and database of University and Hospital Trust of Verona.

The ownership of the data will only be referred to the Principal Investigator (PI) of the project.

TIMELINE OF THE PROJECT Duration of specimen collection: 6 months. This period was estimated on the need to treat patients with COVID-19 immediately Expected duration for the analysis of the data obtained: 2 months. This period has been estimated from the investigators' experience and includes both the analysis of the samples and the statistical analysis of the data obtained.

Total duration of the project: 8 months

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized adults affected by SARS-CoV-2. These patients can be enrolled also for other clinical studies such as off-label or compassionate treatments.

Exclusion Criteria:

* Patients that withdraw informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized adults affected by SARS-CoV-2.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2020-03-26 (Actual); Primary Completion 2020-06-10 (Actual); Study Completion 2020-11-26 (Estimated)

PRIMARY OUTCOMES:
COVID-19 associated immune disorder | 24 hours
  Enumeration of circulating cell subsets by flow cytometry [Cell count/µl]
COVID-19 associated inflammation | 48 hours
  Quantification of plasma levels of different solubles factors (GM-CSF, G-CSF, M-CSF, IFN-γ, IFN-α, IL-1, IL-2, IL-4, IL-5, IL-6, IL-9, IL-10, IL-12 (p70), IL-13, IL-15, IL-17A, IL-17F, IL-17E, IL-21, IL-22, IL-23, IL-27, IL-28A, IL-31, IL-33, IL-34, MIP-3α/CCL20, CCL2, TNF-α, TNF-β, TGFβ) [pg/ml]
Oxygenation | 24 hours
  Ratio of arterial oxygen tension (mmHg) to fraction of inspired oxygen (PaO2/FiO2)
Diagnostic of COVID disease composite | On admission of hospital
  SARS-CoV-2 infection will be tested by PCR using nasopharyngeal swab

SECONDARY OUTCOMES:
Changes at the cytokine pattern | 14 Days
  Quantification of plasma levels of different solubles factors (GM-CSF, G-CSF, M-CSF, IFN-γ, IFN-α, IL-1, IL-2, IL-4, IL-5, IL-6, IL-9, IL-10, IL-12 (p70), IL-13, IL-15, IL-17A, IL-17F, IL-17E, IL-21, IL-22, IL-23, IL-27, IL-28A, IL-31, IL-33, IL-34, MIP-3α/CCL20, CCL2, TNF-α, TNF-β, TGFβ) [pg/ml]
Changes at circulating immune cell composition | 14 Days
  Enumeration of circulating cell subsets by flow cytometry [Cell count/µl]
Intensive Care Unit Admission | Day 7-14
  Proportion of patients with Intensive Care Unit Admission requirement
Length of hospital stay | Day 7-14
  Days of Hospitalization
Clinical Status | Day 7-14
  Clinical status assessed according to the World Health Organization guideline
Mortality | Day 7-14
  Proportion of death patients at days

CONTACTS AND LOCATIONS:
Overall Officials: VINCENZO BRONTE, MD, Principal Investigator — University and Hospital Trust of Verona
Locations (1):
- Azienda Ospedaliera Universitaria Integrata Verona, Verona, Italy

REFERENCES:
- [Background] Moore JB, June CH. Cytokine release syndrome in severe COVID-19. Science. 2020 May 1;368(6490):473-474. doi: 10.1126/science.abb8925. Epub 2020 Apr 17. No abstract available. PMID 32303591
- [Background] Mehta P, McAuley DF, Brown M, Sanchez E, Tattersall RS, Manson JJ; HLH Across Speciality Collaboration, UK. COVID-19: consider cytokine storm syndromes and immunosuppression. Lancet. 2020 Mar 28;395(10229):1033-1034. doi: 10.1016/S0140-6736(20)30628-0. Epub 2020 Mar 16. No abstract available. PMID 32192578
- [Background] Tay MZ, Poh CM, Renia L, MacAry PA, Ng LFP. The trinity of COVID-19: immunity, inflammation and intervention. Nat Rev Immunol. 2020 Jun;20(6):363-374. doi: 10.1038/s41577-020-0311-8. Epub 2020 Apr 28. PMID 32346093
- [Background] Wen W, Su W, Tang H, Le W, Zhang X, Zheng Y, Liu X, Xie L, Li J, Ye J, Dong L, Cui X, Miao Y, Wang D, Dong J, Xiao C, Chen W, Wang H. Immune cell profiling of COVID-19 patients in the recovery stage by single-cell sequencing. Cell Discov. 2020 May 4;6:31. doi: 10.1038/s41421-020-0168-9. eCollection 2020. PMID 32377375
- [Background] Merad M, Martin JC. Pathological inflammation in patients with COVID-19: a key role for monocytes and macrophages. Nat Rev Immunol. 2020 Jun;20(6):355-362. doi: 10.1038/s41577-020-0331-4. Epub 2020 May 6. PMID 32376901
- [Background] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- [Derived] Bronte V, Ugel S, Tinazzi E, Vella A, De Sanctis F, Cane S, Batani V, Trovato R, Fiore A, Petrova V, Hofer F, Barouni RM, Musiu C, Caligola S, Pinton L, Torroni L, Polati E, Donadello K, Friso S, Pizzolo F, Iezzi M, Facciotti F, Pelicci PG, Righetti D, Bazzoni P, Rampudda M, Comel A, Mosaner W, Lunardi C, Olivieri O. Baricitinib restrains the immune dysregulation in patients with severe COVID-19. J Clin Invest. 2020 Dec 1;130(12):6409-6416. doi: 10.1172/JCI141772. PMID 32809969